CLINICAL TRIAL: NCT06629636
Title: Investigate the Efficacy of Using NMN to Improve Embryo Development Capacity and IVF Success Rate in Patients Who Have Experienced IVF Failures.
Brief Title: Investigate the Efficacy of Using NMN to Improve Embryo Development Capacity.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sunkaky Medical Cooperation (Industry)
Collaborators: Abinopharm, Inc (Network); Aba Chemicals Co Ltd (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: IVFJapan202402
Record Dates: First submitted 2024-10-02; First posted 2024-10-08 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-10

CONDITIONS: Repeated IVF Failure; Female Infertility
Keywords: IVF failure; NMN; Female Infertility; Japan; Oocyte Mitochondria; Anti aging
MeSH Terms: conditions — Infertility, Female

STUDY DESIGN:
Intervention Model Description: Dietary Supplement: NMN intervention NMN capsules (total of 900mg/day) for 8 weeks, NMN capsules (total of 900mg/day) for 8 weeks Placebo Comparator: Placebo intervention
  Placebo NMN-free placebo capsules for 8 weeks Other:
  Placebo, for 8 weeks
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- NMN intervention (Active Comparator): NMN capsules (total of 900mg/day) for 8 weeks
  Interventions: Dietary Supplement: NMN capsule
- Placebo intervention (Placebo Comparator): NMN-free placebo capsules for 8 weeks
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: NMN capsule — Total of 900mg/day for 8 weeks
  Arms: NMN intervention
Other: Placebo — NMN-free placebo capsules for 8 weeks
  Arms: Placebo intervention

SUMMARY:
The objective of this study is to investigate the efficacy of NMN supplementation in enhancing embryo developmental capacity and improving IVF success rates in patients experiencing IVF failures.

DETAILED DESCRIPTION:
Reproductive aging is an irreversible process characterized by a decline in oocyte quality, posing a significant challenge to fertility and often leading to unsuccessful outcomes in assisted reproductive technologies. Repeated ART failures can result in substantial burdens for patients, both financially and emotionally. Extensive clinical and preclinical data have established a strong correlation between age-related decline in egg quality and mitochondrial deterioration, resulting in decreased energy production within oocytes. Notably, a reduction in nicotinamide adenine dinucleotide (NAD+ / NADH) concentrations, a crucial redox cofactor and enzyme-substrate essential for energy metabolism, DNA repair, and epigenetic homeostasis, has been observed in various tissues with age.

Recent studies on mice have indicated that Nicotinamide mononucleotide supplementation may mitigate the age-related decline in NAD(P)H levels, enhancing the quality of aged oocytes. This improvement is achieved by promoting both nuclear and cytoplasmic maturation, ensuring euploidy and fertilization competence, ultimately leading to an increased ovulation rate and improved fertility. Moreover, NMN has been shown to restore mitochondrial function in aged oocytes, effectively suppressing the accumulation of reactive oxygen species and DNA damage, and subsequently reducing apoptosis.

Clinical studies have further corroborated the safety and tolerability of NMN supplementation, with daily oral doses of up to 900 mg demonstrating an increase in blood NAD concentrations. Furthermore, research suggests that a daily oral dose of 900 mg maximizes clinical efficacy, as evidenced by blood NAD concentration and physical performance.

This study adopts a triple-blind, randomized, placebo-controlled, prospective pilot study design. This prospective study aims to evaluate the effects of dietary supplementation with 900mg of NMN on ART outcomes in individuals experiencing in vitro fertilization failures attributed to compromised oocyte and embryo quality.

ELIGIBILITY:
Inclusion Criteria:

* Agree to participate in the study
* 32-42 years old
* Having at least one previous embryo implantation failure
* History of low Embryo quality at day3 or day5 (according to Veeck's and Gardner's Criteria)
* No major uterine or ovarian abnormalities
* BMI level 18-25kg/m2

Exclusion Criteria:

* Ovarian endometriosis with Chocolate cysts (AFS type 3 and 4)
* Patients who have taken different supplements such as coenzyme Q10, vitamin E, carnitine,niacin, nicotinamide, or other vitamin B3-related etc. within the previous month
* Any medical contraindication of oocyte retrieval or subsequent procedures
* Couples where the husband presents with severe sperm abnormalities
* Couples where the husband presents <5 million/mL motile sperm
* Uterine structural anomalies
* Polycystic ovaries
* Premature ovarian failure
* Individuals who need regular medication to treat chronic diseases such as diabetes, hypertension, gout, hyperuricemia, etc.
* Individuals who need drug treatment for any mental illness such as epilepsy and depression.
* Individuals who suffer from infectious diseases such as hepatitis B, active tuberculosis, AIDS, etc.
* Cancer patients or receiving chemo/radiotherapy treatment within the past 3 years.

Ages: 32 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-08-20 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Embryo development rate | Up to 8 weeks post-intervention
  Analyze and compare the transferable embryo rate per zygote on day 3 in between NMN and placebo intervention groups.
Changes in metabolic status | Up to 8 weeks post-intervention
  Analyze and compare the NAD+/NADH level in serum and follicular fluid in both NMN and placebo groups
Clinical pregnancy rate | Up to 12months post-intervention
  Compare ongoing clinical pregnancy rates between NMN and placebo groups
Embryo development rate | Up to 8 weeks post-intervention
  Analyze and compare the quality of embryos on day 3, 5 or 6 between two groups
Embryo development rate | Up to 8 weeks post-intervention
  Analyze and compare the rate of blastocyst development on day 5 and 6 in between two groups

SECONDARY OUTCOMES:
Live Birth rates | Up to 24 months post-intervention
  Compare live Birth rate following the intervention in both groups
Endocrine hormones including AMH | Up to 8 weeks post-intervention
  Changes in endocrine hormones including AMH levels in serum after the interventions.
Average egg retrieval capacity per person | Up to 8 weeks post-intervention
  Compare the number of antral follicles in each ovary will be determined using transvaginal ultrasonography in both groups.
Additional in vitro fertilization - outcome indicators | Up to 8 weeks post-intervention
  Number of average recruited MII oocytes in both groups
Chemical pregnancy rate | Up to 12months post-intervention
  Compare the chemical pregnancy rates between the two groups.
Pregnancy complication | Up to 24 months post-intervention
  Rate of pregnancy complication in both groups
Abortion rate | Up to 24 months post-intervention
  Compare the abortion rates in both groups
Additional in vitro fertilization - outcome indicators | Up to 8 weeks post-intervention
  Compare the rate of fertilization in between two groups
Additional in vitro fertilization - outcome indicators | Up to 8 weeks post-intervention
  Rate of abnormal fertilization in both groups
Additional in vitro fertilization - outcome indicators | Up to 8 weeks post-intervention
  The rate of non-transferable embryos in both groups

CONTACTS AND LOCATIONS:
Overall Officials: Yoshiharu M., Yoshiharu Morimoto, MD, PhD, Principal Investigator — Sankaky Medical Corporation; Naoharu M., Naoharu Yoshiharu, MD, Study Director — Sankaky Medical Corporation
Locations (1):
- IVF Namba Clinic, Sankaky Medical Corporation, Osaka, Osaka, Japan

IPD SHARING:
Plan to Share IPD: No
The confidentiality of patients' information is strictly maintained.

REFERENCES:
- [Background] Huang H. A Multicentre, Randomised, Double Blind, Parallel Design, Placebo Controlled Study to Evaluate the Efficacy and Safety of Uthever (NMN Supplement), an Orally Administered Supplementation in Middle Aged and Older Adults. Front Aging. 2022 May 5;3:851698. doi: 10.3389/fragi.2022.851698. eCollection 2022. PMID 35821806
- [Background] Yi L, Maier AB, Tao R, Lin Z, Vaidya A, Pendse S, Thasma S, Andhalkar N, Avhad G, Kumbhar V. The efficacy and safety of beta-nicotinamide mononucleotide (NMN) supplementation in healthy middle-aged adults: a randomized, multicenter, double-blind, placebo-controlled, parallel-group, dose-dependent clinical trial. Geroscience. 2023 Feb;45(1):29-43. doi: 10.1007/s11357-022-00705-1. Epub 2022 Dec 8. PMID 36482258
- [Background] Miao Y, Cui Z, Gao Q, Rui R, Xiong B. Nicotinamide Mononucleotide Supplementation Reverses the Declining Quality of Maternally Aged Oocytes. Cell Rep. 2020 Aug 4;32(5):107987. doi: 10.1016/j.celrep.2020.107987. PMID 32755581
- [Background] Bertoldo MJ, Listijono DR, Ho WJ, Riepsamen AH, Goss DM, Richani D, Jin XL, Mahbub S, Campbell JM, Habibalahi A, Loh WN, Youngson NA, Maniam J, Wong ASA, Selesniemi K, Bustamante S, Li C, Zhao Y, Marinova MB, Kim LJ, Lau L, Wu RM, Mikolaizak AS, Araki T, Le Couteur DG, Turner N, Morris MJ, Walters KA, Goldys E, O'Neill C, Gilchrist RB, Sinclair DA, Homer HA, Wu LE. NAD+ Repletion Rescues Female Fertility during Reproductive Aging. Cell Rep. 2020 Feb 11;30(6):1670-1681.e7. doi: 10.1016/j.celrep.2020.01.058. PMID 32049001
- [Background] Schultz MB, Sinclair DA. Why NAD(+) Declines during Aging: It's Destroyed. Cell Metab. 2016 Jun 14;23(6):965-966. doi: 10.1016/j.cmet.2016.05.022. PMID 27304496
- [Background] Bentov Y, Yavorska T, Esfandiari N, Jurisicova A, Casper RF. The contribution of mitochondrial function to reproductive aging. J Assist Reprod Genet. 2011 Sep;28(9):773-83. doi: 10.1007/s10815-011-9588-7. Epub 2011 May 27. PMID 21617930
- [Background] Hashimoto S, Morimoto Y. Mitochondrial function of human embryo: Decline in their quality with maternal aging. Reprod Med Biol. 2022 Dec 21;21(1):e12491. doi: 10.1002/rmb2.12491. eCollection 2022 Jan-Dec. PMID 36570768